CLINICAL TRIAL: NCT06097897
Title: Evaluation of a Non-Invasive Imaging Device for the Acquisition of Imaging Data of Vitreous Opacities in Human Eyes
Brief Title: Imaging of Vitreous Opacities in Human Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PulseMedica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SVO-IDFIH001
Record Dates: First submitted 2023-09-26; First posted 2023-10-24 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Floaters; Vitreous Opacities
MeSH Terms: conditions — vitreous floaters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imaging using the SVO-ID (Experimental): Patients will have their eyes imaged with the SVO-ID as part of a study visit.
  Interventions: Device: SVO-ID

INTERVENTIONS:
Device: SVO-ID — Combined scanning laser ophthalmoscope (SLO) and optical coherence tomography (OCT) for imaging of the eye

SUMMARY:
Vitreous opacities (VOs), commonly known as floaters, are dark spots that appear in, and may float across your vision. Presently, there is a lack of available data in the literature regarding VOs. This study aims to obtain imaging data of VOs in the population to build an imaging database of VOs to learn more about them.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* SVO-related symptoms in vision
* Clear ocular media, to allow a clear view of the vitreous for the SVO-ID

Exclusion Criteria:

* Presence of vitreous hemorrhage
* Cataract Grade 3 and above
* Opacification of lens, cornea, or vitreous
* Diagnosis of narrow-angle glaucoma
* Refractive error is outside the range of -6D to +3D
* Astigmatism is outside the range of +/- 2D of cylinder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Successful capture of SLO and OCT imaging data of SVOs for algorithm development | Through study completion, an average of one year
  Successful collection of SLO and OCT imaging data

SECONDARY OUTCOMES:
Collection of patient-reported symptoms | Through study completion, an average of one year
  Patient feedback regarding symptoms related to SVOs being imaged

CONTACTS AND LOCATIONS:
Locations (1):
- Panama Eye Center, Panama City, Panama